CLINICAL TRIAL: NCT04573842
Title: Ultrasound Assessment of the Subclavian Vein for Predicting Hypotension in Children After Anaesthesia Induction
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Jacob Karlsson, Principal Investigator, Karolinska Institutet
Other Study IDs: KarolinskaSCV
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia Complication; Hypotension on Induction; Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Ultrasound assessment of SCV — An ultrasound examination of the SCV will be performed before anesthesia induction. Apart from this, the protocol does not differ at all from the ordinary fashion

SUMMARY:
Intra operative hypotension is a risk factor in pediatric anesthesia (McCann ME et al.Pediatr Anesth 2014; 24: 68-73). In summary, the study aims at examine if ultrasound assessment of the diameter and collapsibility index of the subclavian vein is correlated to fasting time and if they are correlated to the degree of hypotension seen post anesthesia induction in children undergoing general anesthesia.

DETAILED DESCRIPTION:
Background: Intra operative hypotension is a risk factor in pediatric anesthesia (McCann ME et al.Pediatr Anesth 2014; 24: 68-73). Bedside ultrasonic assessment of the inferior vena cava (IVC) and IVC collapsibility index (IVCCI) has been shown to indicate fluid status in both adults and children breathing spontaneously (Marcell Szabó et al. BMC Anesthesiol. 2019; 19: 139., Lei Chen et al.Acad Emerg Med. 2007 Oct;14(10):841-5.). Ultrasound assessment of subclavian vein/axillary vein collapsibility has recently been shown to predict hypotension after induction of general anesthesia in adults (Min Hee Choi et al. Eur J Anaesthesiol 2020; 37:474-481). The inverstigators hypothesized that subclavian vein (SCV) collapsibility index is correlated to fasting time and potentially can be used to predict post induction hypotension in children.

Objective: To examine if ultrasound assessment of the diameter and collapsibility index of the SCV is correlated to fasting time and can be a predictor of post induction hypotension in children undergoing general anesthesia.

Design and setting: Prospective observational study in a day case surgical unit in a tertiary university hospital.

Patients: Children aged 0-18 years ASA 1-2 undergoing anesthesia for day case surgery after written and informed consent from parents is obtained according to local ethical permit. Exclusion criteria: ongoing medication for hypertension.

Measurements and results: Based on previous studies (Min Hee Choi et al. Eur J Anaesthesiol 2020; 37:474-481), a sample size of approximately 80 subjects will be needed. Data on fasting time will be collected after informed and written consent has been obtained. Before the induction of anesthesia, the patients will be breathing spontaneously in a supine position. Noninvasive blood pressure will be recorded. An ultrasound examination of SCV will then be performed on cross section of the vessel both in 2D and M-mode and the minimum and maximum diameters of the SCV will be recorded. Collapsibility index will then be calculated from these data as previously described (Min Hee Choi et al. Eur J Anaesthesiology 2020; 37:474-481). After this, the subjects will undergo anesthesia under which blood pressure will be recorded according to departmental standard as usual. SCV collapsibility index will then be investigated for potential significant correlation with fasting time and percentage decrease in blood pressure from baseline after anesthesia induction and during the surgical preparation phase, before start of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children undergoing anesthesia for day case surgery in the age group newborn to eighteen years.

Exclusion Criteria:

* Ongoing medication for hypertension. ASA status of more than 2.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children aged 0-18 years ASA 1-2 undergoing anesthesia for day case surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-10-07 (Actual)

PRIMARY OUTCOMES:
SCV Collapsibility index correlation to post induction hypotension | 120 minutes
  SCV Collapsibility index correlation to percentage change in non invasive blood pressure from baseline recordings pre anesthesia induction

SECONDARY OUTCOMES:
SCV Collapsibility index correlation to fasting time | 120 min minutes
  SCV Collapsibility index correlation to fasting time in hours

OTHER OUTCOMES:
Fasting time correlation to post induction hypotension | 120 minutes
  percentage change in non invasive blood pressure from baseline recordings pre anesthesia induction

CONTACTS AND LOCATIONS:
Overall Officials: Per-Arne Lönnqvist, Prof, Study Chair — Karolinska University
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No